CLINICAL TRIAL: NCT03409042
Title: Caloric Compensation in Infants
Status: Completed | Type: Observational
Sponsor: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Responsible Party: Sponsor
Other Study IDs: PUNCH 1.1.2 (2015-A00014-45)
Record Dates: First submitted 2018-01-18; First posted 2018-01-24 (Actual); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Self Regulation; Eating Behavior; Infant Behavior
Keywords: Caloric compensation
MeSH Terms: conditions — Self-Control; Feeding Behavior; Infant Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Caloric compensation — The investigators have adapted an established within-subject preload paradigm to assess infant's short term caloric compensation. At each studied age, the measure of caloric compensation required two visits at the laboratory on two non-consecutive days. On the first visit, the infants received a fixed amount of a food preload either low or high in energy density. The order of the two preloads was counterbalanced. After a delay (ranging from several hours in the 3-4 months old infants to 25 min in 10.5- and 14.5-month-old infants), the infants were served an ad libitum meal. Weight intakes (g) were assessed by weighing each bottle/bowl before and after consumption.

SUMMARY:
The aim of this study is, first, to describe the evolution of the caloric compensation ability in infants from 3 to 15 months old and, secondly, to assess the links between changes in the caloric compensation ability and the individual characteristics (adiposity, age, gender, infant's eating behavior) and maternal feeding practices.

Three series of measurements of caloric compensation abitlity were conducted: at 3-4 months old, at 10.5 months old and at 14.5 months old in the laboratory.

In this study, a preload paradigm usually employed in children and adults to measure the caloric compensation ability was adapted to infants below 15 months old. The maternal eating behavior and their feeding practices were measured by questionnaires. The infants' height and weight were measured at the laboratory by trained experimenters.

ELIGIBILITY:
Inclusion Criteria:

* no chronic health problem or food allergies
* not having been fed with hydrolysate formula
* gestational age ≥ 37 weeks
* born weight ≥ 2.5kg
* without having being tube fed at any moment

Exclusion Criteria:

* infants from diabetic mothers
* infants from mothers having celiac disease
* infants from minor parents (<18 years old) were excluded

Ages: 3 Months to 11 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Recruitment was conducted using leaflets distributed in health professionals' consulting rooms, an internal database (Chemosens Platform's PanelSens, CNIL n°1148039) and with the help of a recruitment agency.
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
COMPX score | one week
  Based on intake data, Energy Intakes (EI) were calculated according to caloric composition of the offered foods from the manufacturers. From the EI data, a COMPX score was calculated at each studied age by dividing the difference in EI from meals by the difference in EI from preloads (presented as a percentage). A COMPX score of 100% reflects a perfect caloric compensation.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Birch, L.L. and M. Deysher, Conditioned and unconditioned caloric compensation: evidence for self regulation of food intake in young children. Learning and Motivation, 1985. 16: p. 341-355.
- [Derived] Brugailleres P, Chabanet C, Issanchou S, Schwartz C. Caloric compensation ability around the age of 1 year: Interplay with the caregiver-infant mealtime interaction and infant appetitive traits. Appetite. 2019 Nov 1;142:104382. doi: 10.1016/j.appet.2019.104382. Epub 2019 Jul 23. PMID 31348973
- [Derived] Brugailleres P, Issanchou S, Nicklaus S, Chabanet C, Schwartz C. Caloric compensation in infants: developmental changes around the age of 1 year and associations with anthropometric measurements up to 2 years. Am J Clin Nutr. 2019 May 1;109(5):1344-1352. doi: 10.1093/ajcn/nqy357. PMID 30997507